CLINICAL TRIAL: NCT00269997
Title: The Effect of Subcutaneous r-HuEPO in Patients With Chronic Anemia Secondary to Cisplatin Chemotherapy
Brief Title: A Study to Evaluate the Safety and Effectiveness of Epoetin Alfa Versus Placebo in Patients With Persistent Anemia as a Result of Cancer Treatment With Cisplatin, a Platinum-containing Chemotherapy Drug
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005839
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Neoplasms
Keywords: Anemia; chemotherapy; epoetin alfa; epogen; erythropoietin; neoplasms; cancer
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of epoetin alfa versus placebo in the treatment of persistent anemia caused by advanced cancer and aggressive cisplatin chemotherapy. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Patients undergoing treatment with cisplatin-containing chemotherapy frequently develop significant anemia (hemoglobin <= 10.5 grams/deciliter). Agents that can increase the amount of hemoglobin in cancer patients undergoing treatment with cisplatin-containing cyclic chemotherapy may improve the patients' reduced physical strength and reduced stamina resulting from anemia, increase the patients' ability to continue chemotherapy, and improve the patients' overall qualify of life. Epoetin alfa is a genetically engineered form of a natural hormone (erythropoietin) that is used to treat anemia by stimulating red blood cell production. This is a randomized, double-blind, placebo-controlled, parallel group, multicenter study. This study evaluates the safety and effectiveness of epoetin alfa in treating patients who develop persistent anemia as a result of treatment with aggressive cisplatin-containing cyclic chemotherapy (every 3 to 4 weeks) for any cancer type (except rapid and severe onset of leukemias and malignancies of the bone marrow and spleen). The study consists of a <= 7 day screening period when patients' eligibility is determined, a 12-week double-blind treatment period, and an optional open-label treatment period. Eligible patients will be randomly assigned to one of two treatment groups: epoetin alfa 150 units/kilogram or a comparable volume of placebo, given by injection beneath the skin. Patients will be treated with study medication 3 times weekly for 12 weeks. Two of the 3 weekly doses of study medication may be self-administered by the patient at home; the patient is visited by a health professional at least once weekly to administer the other dose(s). The dose of study medication may be increased or decreased at the discretion of the physician, based on the results of blood tests. Depending on the patient's chemotherapy cycle, he or she will return to the study site every 3 or 4 weeks for administration of study medication. During the open-label treatment period, patients who choose to continue will receive 3 injections per week of epoetin alfa under the skin, until the completion of his or her chemotherapy treatments. Safety evaluations, including laboratory tests, vital signs, reporting of adverse events, physical examination, and electrocardiograms, are performed throughout the study. Effectiveness of the study drug will be determined by the number of transfusions patients require and by changes in blood test results (hemoglobin, hematocrit, and immature red blood cells) from before the start of the study to the end of the study. The study hypothesis is that epoetin alfa will, more effectively than placebo, stimulate adequate production of red blood cells to elevate the hemoglobin level in cancer patients who are anemic as a result of undergoing treatment with aggressive cisplatin-containing cyclic chemotherapy. Double-blind: Epoetin alfa 150 units/kilogram, or matching volume of placebo, injected beneath the skin 3 times weekly for 12 weeks. Open-label: Epoetin alfa at the dose received at the end of the double-blind study injected beneath the skin 3 times weekly for any remaining cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer (except for rapid onset of severe leukemia and malignancies of the bone marrow and spleen) and having anemia resulting from cisplatin-containing chemotherapy
* receiving cyclic chemotherapy for <=5 consecutive days every 3 or 4 weeks (for 3 cycles of chemotherapy)
* Performance score of 0, 1, 2, or 3 (grades assessing patients' ability to perform daily activities)
* having a life expectancy of at least 3 months
* having a hemoglobin level <= 10.5 grams/deciliter, and signs and symptoms of physical stability for 1 month before the study (based on physical examination including vital signs, weight, and electrocardiogram)
* with an ability to administer self-injections

Exclusion Criteria:

* Patients with a history of any blood disease
* having signs and symptoms of significant disease/dysfunction not caused by the underlying cancer
* receiving radiation therapy or surgery to decrease the number of cancer cells within 30 days before the start of the study
* having a sudden and severe onset of illness within 7 days before the start of the study
* having cancer that has spread to the brain, a history of seizures, uncontrolled high blood pressure, or an iron, folate, or vitamin B12 deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Study Completion 1990-07 (Actual)

PRIMARY OUTCOMES:
Number of transfusions required; Changes in hemoglobin, hematocrit, and reticulocyte (immature red blood cells) levels from before the study to the end of the study

SECONDARY OUTCOMES:
Quality of life assessment; Physician's global evaluation; Performance score (ability to perform daily activities); Assessment of safety (laboratory tests, vital signs, and adverse events) from before the study to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study to evaluate the safety and effectiveness of epoetin alfa given by injection beneath the skin to patients with persistent anemia as a result of cancer treatment with cisplatin, a platinum-containing anti-cancer drug — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=672&filename=CR005839_CSR.pdf